CLINICAL TRIAL: NCT04237051
Title: Knowledge, Attitude and Practice (KAP) Among Fifth Year Undergraduate Dental Students, Cairo University Towards Ergonomics: Cross -Sectional Study
Brief Title: Knowledge, Attitude and Practice Among Undergraduate Dental Students, Cairo University Towards Ergonomics
Status: Completed | Type: Observational
Sponsor: Wessam Maher Gomaa Tag El-Dein (Other)
Responsible Party: Sponsor-Investigator, Wessam Maher Gomaa Tag El-Dein, postgraduate student in faculty of dentistry cairo university, Cairo University
Organization: Cairo University (Other)
Other Study IDs: CEBD-CU-2020-01-18
Record Dates: First submitted 2020-01-17; First posted 2020-01-22 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-01

CONDITIONS: Knowledge, Attitudes, Practice
Keywords: knowledge; attitude; practice; KAP; ergonomics; dental ergonomics
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
this study will evaluate knowledge, attitude, and practice of fifth-year dental students Cairo university toward ergonomics

DETAILED DESCRIPTION:
Ergonomic is the study of people and their working environment. Ergonomic consequently is the science concerned with designing products and procedures to maximize efficiency and safety.

The world health organization defines Musculoskeletal disorder (MSD) as "a disorder of the muscles Tendons, joints, intervertebral discs, Peripheral nerves, and vascular system''.

The musculoskeletal disorders are common among medical professionals, and especially dentists and dental hygienists, because of the prevalence of different postures in dental procedures, prolonged stature, unsupported sitting, griping smaller and thin instruments for a longer time and limited access during dental procedures.

Musculoskeletal disorder (MSD) affect muscle, joints, tendons, ligaments, and nerves and caused by work itself or by working environment. It has been reported that back pain is the most common followed by neck pain and shoulder pain. If early signs and symptoms are noted, with the understanding of mechanisms of progression of the disease, MSDs can be prevented at earlier stage.

(Gupta et al., 2014), state some signs and symptoms of MSD on dentists:

Signs of MSDs:

* Decreased range of motion.
* Loss of normal sensation.
* Decreased grip strength.
* Loss of normal movement.
* Loss of coordination.

Symptoms of MSDs:

* Excessive fatigue in the shoulders and neck.
* Tingling, burning or other pain in arms.
* Weak grip, cramping of hands.
* Numbness in fingers and hands.
* Clumsiness and dropping of objects.
* Hypersensitivity in hands and fingers.

Goals of Ergonomics according to (Pendyala and Karunakar, 2014) :

* Prevention of work-related musculoskeletal disorders and conditions which might lead to it.
* Increasing safety and productivity.
* Enhanced performance by eliminating unnecessary effort.
* Improving the standard of care to the patient.

So this study is conducted to assess the knowledge, attitude, and practice (KAP) among fifth-year undergraduate dental students, Cairo University towards Ergonomics

ELIGIBILITY:
Inclusion Criteria:

* Fifth-year undergraduate dental students, Cairo University at the time of the study

Exclusion Criteria:

* Refusal to participate

Ages: 21 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: all fifth year dental students at Cairo university
Sampling Method: Non-Probability Sample
Enrollment: 374 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
knowledge,attitude,and practice toward ergonomics | 2 months using percentage scale from 0%-100% where higher score means better outcome
  self reporting questionnaire for knowledge,attitude,and practice toward ergonomics

CONTACTS AND LOCATIONS:
Overall Officials: hassan ahmed, Principal Investigator — center of evidence based dentistry
Locations (1):
- Wessam Maher, Cairo, Mokatam, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
due to financial issue